CLINICAL TRIAL: NCT02090491
Title: MENTIS Personal Health Record Rapid Pilot Research Deployment and Evaluation
Status: Completed | Type: Observational
Sponsor: Northeastern University (Other)
Responsible Party: Sponsor
Other Study IDs: Janssen Research & Development
Record Dates: First submitted 2013-11-01; First posted 2014-03-18 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Autism
Keywords: autism
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Autism Spectrum Disorder (ASD) is a collection of complex neurodevelopmental disorders characterized by qualitative impairments in socialization, communication, and circumscribed interests, including stereotypical behavior patterns and behavioral rigidity to changes in routines (American Psychiatric Association, 1994). ASD is the fastest growing pervasive developmental disorder of childhood, currently estimated to affect 1 in 88 school age children (Baio, 2012). ASD typically manifests in infancy and persist throughout the lifespan. There is no known cause or cure for ASD, yet structured behavioral interventions and medications can enhance developmental outcomes. ASD has a profound impact on families and often result in enormous emotional and financial costs. Recent estimates suggest that societal costs in the US to care for all individuals diagnosed each year over their lifetime approaches $35 billion (Ganz, 2007).

Janssen Research & Development is building a comprehensive digital platform (MENTIS) to optimize and enhance development of novel medicines and track outcomes in individuals with ASD. The MENTIS platform contains several core components, including: (1) An electronic personal healthcare record, designed specifically for individuals with ASD and their caregivers (parents, teachers, healthcare providers); (2) Integrated physiological and physical activity biosensors designed to objectively assess outcomes important in ASD, and; (3) A de-identified research data warehouse with analytic tools to better measure outcomes, assist with sub-population identification, and identify algorithms for diagnosis and treatment response detection.

The MENTIS platform is currently being designed, developed, and prepared for testing. During this process it is highly desirable to conduct feasibility and usability research with a sample of the target population to identify important system components and features, optimize design, and reduce redundancy in software development and research time. The rapid pilot study described herein is proposed to gather incipient feedback on select MENTIS system components and features from stakeholders who support individuals with ASD in a clinical setting. This pilot research will help evaluate both how well current MENTIS system features work in an applied setting and inform future directions for MENTIS platform development.

ELIGIBILITY:
Inclusion Criteria:

Student Participants:

* Meet standard classroom selection criteria of age, gender, intellectual ability, communication ability and behavioral characteristics (frequency and duration of maladaptive behaviors).
* Be enrolled at Center for Discovery, have a Behavioral Intervention Plan (BIP), and an Individualized Education Plan (IEP).
* Have a diagnosis of autism.
* Be between the ages of 5 and 21 years, inclusive.
* Tolerate wearing physiological wrist, ankle, and chest monitors.

Residential and School Staff:

* Employed at The Center for Discovery.
* Meet Center for Discovery requirements for working with students in the classroom or residence and have experience in teaching or intervening with students who exhibit maladaptive behaviors.
* Willing to consent to add data to the system via the supplied tablet for the duration of the study.
* Willing to consent to participate in either focus groups or individual interviews about their experience of using the system and to be video recorded doing so.

Parent Participants:

* Be the parent or legal guardian of one of the 20 students enrolled in the study.
* Willing to consent to add data to the system via the supplied tablet for the duration of the study.
* Willing to consent to participate in either focus groups or individual interviews about their experience using the system and to be video recorded doing so.

Exclusion Criteria:

Student Participants:

* Younger than 5 years at the start of the school year.
* Not reach the age of 21 years prior to the end of the school year during which the study will take place.
* Not enrolled at Center for Discovery.
* Do not tolerate wearing physiological monitors after repeated trials of modeling, desensitization, shaping, and reinforcement.

Residential and School Staff:

* Have not been employed for at least one year prior to participating in the study.
* Do not consent to adding data.
* Do not consent to participant in focus groups or interviews.
* Do not consent to being recorded during focus groups or interviews.

Parent Participants:

* Are not the parent or legal guardian of one of the student enrolled.
* Do not consent to participate in either focus groups of individual interviews about their experience using the system and to be video recorded doing so.

Ages: 5 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Group 1: Six (6) students from the Discovery School and their respective support staff. Inclusion criteria include a diagnosis of ASD and enrollment in the Discovery School due to frequently observed challenging behaviors. Reporters will include: 2 teachers, HCP and parent/guardian.
  Group 2: Fourteen (14) students receiving services from Center for Discovery (but outside the Discovery School), their respective support staff, and, for those who live at home, their parents. Inclusion criteria includes a diagnosis of ASD, seven (7) students who reside in a CfD provided campus home, and seven (7) students who reside in the local community with their parents. Reporters will include: 2 teachers, HCP, residential staff and parents.
  Stakeholders: Healthcare professionals, classroom teachers, residential staff, and parents who support students with ASD in Groups 1 and 2 above.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Self-Report | 6 months
  Summary of data from all data collection cycles (includes Stakeholder entered data, biosensor data and passive system usage data) in aggregate and raw, de-identified dataset with both qualitative and quantitative information:
  * Qualitative and quantitative data from Exit Interviews
  * System usage data;
  * Pre-post summary,
  * case examples,
  * de-identified video examples,
  * testimonials,
  * overall results.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew S Goodwin, PhD, Principal Investigator — Northeastern University
Locations (1):
- Center for Discovery, Harris, New York, United States